CLINICAL TRIAL: NCT06333002
Title: Developing an Optimal Machine Learning Model to Predict ICU Outcome in Patients With Acute Hypoxemic Respiratory Failure
Brief Title: Machine Learning Model to Predict Outcome in Acute Hypoxemic Respiratory Failure
Acronym: MEMORIAL
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Jesus Villar, principal investigator, Dr. Negrin University Hospital
Other Study IDs: PI24/00325
Record Dates: First submitted 2024-03-19; First posted 2024-03-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: outcome; mechanical ventilation; machine learning
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Logistic Models

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Derivation cohort: It will contain 800 patients randomly selected (1,000 patients with AHRF)
  Interventions: Other: machine learning analysis
- Validation cohort: It will contain 200 patients randomly selected (20% of 1000 patients with AHRF
  Interventions: Other: machine learning analysis
- Confirmatory cohort: It will contain the remaining 241 patients randomply selected (por external validation)
  Interventions: Other: machine learning analysis

INTERVENTIONS:
Other: machine learning analysis — We will use robust machine learning approaches, such as Random Forest, Extreme Gradient Boosting, Support Vector Machine and Multilayer Perceptron.
  Other Names: Logistic regression, cross validation, and area under the ROC curves

SUMMARY:
Acute hypoxemic respiratory failure (AHRF) is the most common cause of admission in the intensive care units (UCIs) worldwide. We will assess the value of machine learning (ML) techniques for early prediction of ICU death in 1,241 patients enrolled in the PANDORA (Prevalence AND Outcome of acute Respiratory fAilure) Study in Spain. The study was registered with ClinicalTrials.gov (NCT03145974). Our aim is to evaluate the minimum number of variables models using logistic regression and four supervised ML algorithms: Random Forest, Extreme Gradient Boosting, Support Vector Machine and Multilayer Perceptron.

DETAILED DESCRIPTION:
Acute hypoxemic respiratory failure (AHRF) is the most common cause of admission in the intensive care units (UCIs) worldwide. We will assess the value of machine learning (ML) techniques for early prediction of ICU death in AHRF patients on mechanical ventilation (MV). Few studies have investigated the prediction of mortality in patients with AHRF.

For model development, the investigators will extract data for the first 2 days after diagnosis of AHRF from patients included in the de-identified database of the PANDORA cohort. We had a database with 2,000,000 anonymized and dissociated demographics and clinical, data from 1,241 patients with AHRF enrolled in our PANDORA cohort (Prevalence AND Outcome of acute Respiratory fAilure) from 22 Spanish hospitals and coordinated by the principal investigator (JV). The investigators will follow the Transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD) guidelines for model prediction. We will screen collected variables employing a genetic algorithm variable selection method to achieve parsimony. We evaluated the minimum number of variables models using logistic regression and 4 supervised ML algorithms: Random Forest, Extreme Gradient Boosting, Support Vector Machine and Multilayer Perceptron. We will use a 5-fold cross-validation in the dataset of 1,000 patients selected randomly in training data (80%) and testing data (20%). For external validation, we will use the remaining 241 patients.

ELIGIBILITY:
Inclusion Criteria:

* endotracheal intubation plus mechanical ventilation (MV)
* PaO2/FiO2 ratio ≤300 mmHg under MV with positive end-expiratory pressure (PEEP) ≥5 cmH2O and FiO2 ≥0.3.

Exclusion Criteria:

* Post-operative patients ventilated <24 h
* Brain death patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: De-identified dataset inclusing 1,241 mechanically ventilated patients with acute hypoxemic respiratory failure admitted consecutively in a network of Spanish ICUs.
Sampling Method: Non-Probability Sample
Enrollment: 1241 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | up to 100 weeks (from inclusion to death or diascharge from intensive care unit
  death in the intensive care unit

SECONDARY OUTCOMES:
MV duration | up to 100 weeks (from inclusion to extubation)
  duration of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Villar, MD, PhD, Principal Investigator — Fundación Canaria Instituto de Investigación Sanitaria de Canarias
Locations (8):
- Spain (8):
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Virgen de La Luz, Cuenca
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Universitario NS de Candelaria, Santa Cruz de Tenerife
  - Hospital Cinico de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No